CLINICAL TRIAL: NCT07289724
Title: MUltiple Sclerosis, How to Instigate Care integrAtion Across nationaL Contexts Via patIentS' Engagement?
Brief Title: How to Develop the Highest Possible Leading-edge Interdisciplinary Care Model for People With MS, That Will be Relevant to All Stakeholders and Declinable to Different Local Contexts With the Ultimate Goal of Ensuring the Highest Level of Quality of Care in MS.
Acronym: MUSICALISE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250160
Record Dates: First submitted 2025-09-30; First posted 2025-12-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; care pathway; coordination of care; multiple sclerosis care units
MeSH Terms: conditions — Multiple Sclerosis | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient: Patient with MS
  Interventions: Other: Focus group; Other: individual interview
- Healthcare professional: Healthcare professional working with MS patients;
  Interventions: Other: Focus group; Other: individual interview
- Carer: Carer for someone with MS
  Interventions: Other: Focus group; Other: individual interview

INTERVENTIONS:
Other: Focus group — With regard to focus groups, these group interviews will take place at specialist centres. Three CRC centres have agreed to host them on their premises. Groups of 6 to 8 people will be invited, the average duration of half a day, or approximately 3½ hours, including welcome and a break. In each of the three approved expert centres, there will be a group composed solely of patients and carers, followed by a group composed of healthcare professionals who are experts in MS, and finally a mixed group (i.e. three FG sessions and therefore three different half-days in each centre three centres).
Other: individual interview — The semi-structured individual interview contains topics that have been thought out in advance, but their form and order are left to the flow of the interview. This type of interview takes the form of a conversation in order to reduce the artificial nature of the exchange. It is an interaction between the researcher and the interviewee whose experience is of direct interest to the research being conducted.

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory, demyelinating and degenerative disease of the central nervous system. It is currently not curable, although several disease-modifying treatments (DMT) reduce the occurrence of relapses and slow disability progression. It affects about 2.8 million persons worldwide (1 million in Europe) with 3 women per 1 man. MS usually starts between 20 and 40 years old, and most people live with the disease for several decades, as life expectancy is reduced by 6-13 years compared to general population. Disease courses are highly heterogeneous and unpredictable at individual level. MS may lead to limited walking abilities but also to invisible symptoms: cognitive dysfunction, pain, bladder dysfunction, and fatigue. This results in a very high burden on affected persons, their families and society. Overall costs among 30 European countries were evaluated in 2010 to 14.559 million euros.

The chronic nature of MS implies a high level of use of health services during the entire life span. MS-specific therapeutic options have undergone extensive development since the 2000s, as well as the understanding of the usefulness of comprehensive MS care. The usual core component of MS care is the neurologist/general practitioner (GP) dyad, and only neurologists are allowed to prescribe MS-specific DMT. With the expanding therapeutic area (and the required strategies to prevent and minimize the risks of adverse events) combined with the heterogeneity of the course and the symptoms, it is more and more difficult for a single physician to acquire and maintain the expertise necessary to comply with gold standard care. Patients may also need referrals to other specialists (physiotherapists, neuropsychologists, psychiatrists, occupational therapists…) depending on their needs. They sometimes use the terms "labyrinth" or "obstacle course" to describe the complex, non-linear, multi-professionals' pathway they are facing.

In the past years, the concept of multidisciplinary MSCU emerged as an organisational innovation, and structures were established at different scales in several countries. These teams available in a single place provide the high level of expertise needed for complex cases or specific steps of the care process. They also dispense formalized diagnostic procedures, protocols for initiation and follow-up of DMT. Their organisation can vary across regions and healthcare systems and needs to be balanced with clinical practice according to local conditions. Thus, there are about 2450 neurologists (67% in public hospitals, 33% private practice) in France, and 23 MS expert centres were labeled by the Ministry of Health in 2017 (one per region, systematically in university public hospitals). In Italy, there are approximately 8000 neurologists and 240 MS centres of varying size, often located within neurology departments in public hospitals. The ability to coordinate interdisciplinary care in each MS centre depends on the capacity and quality of the local health and social care system. The presence of such a new actor in MS management leads to new questions regarding its role and place in the pre-existing system, and how the previous actors (mainly general neurologists, GP, people with MS) accept or use it. To date, little is known on the impact of MSCU on integrated care and personalized approach. Therefore, it is crucial to understand how key stakeholders, such as health professionals, payers and people affected by MS perceive this new and innovative element of the care pathway.

DETAILED DESCRIPTION:
MUSICALISE will help to better understand what is covered by the MSCU concept and what its impacts are in terms of quality of care and care integration. Case studies will be performed in France and Italy, as these two countries have implemented MSCU in different ways. Indeed, the French Ministry of Health has chosen to label regional MS-expert centers, i.e. 23 over the French territory to answer potential needs of about 120,000 patients with MS. In Italy, a different strategy was operated with more than 240 MS centres across the country and around 87% of people with MS (of about 137,000) receive care in these centres. Such choices imply differential use of MSCU, and possibly differential impacts, which will be assessed and measured in the present project. In-depth analysis will be performed in these two pilot countries, with comparisons both between and within countries. In addition, the European Charcot Foundation, collaborator in this project, is currently performing an international survey on MSCU and their implementation in different countries. The data gathered with this survey will be made available to us and will reinforce our understanding on how MS care is delivered and received in different contexts and different countries. This additional data provision will allow us to extend the analysis and leverage our propositions.

The overall objective of MUSICALISE is to develop the highest possible leading-edge interdisciplinary care model that optimizes the integration of care for people living with MS, and therefore the overall quality of care. There is a crucial need for advancing research about MS management and care models, specifying the role and impacts of MSCU to assess its sustainability. Furthermore, the proposed model will be co-constructed to be relevant and declinable in different contexts and answer needs from all the stakeholders (people with and affected by MS, health care providers, and policy makers). To meet this objective, the study will use focus groups and individual interviews.

In that perspective, MUSICALISE has defined 2 specific objectives that involve patients:

* Define the appropriate care pathway based upon the perceptions and experiences of people with MS and that of health care providers involved in MS management. Due to heterogeneity of the disease, it is envisaged to define a "matrix"/journey with the different potential health events (specific to MS or linked to comorbidities) and the appropriate care to provide with the relevant health care providers. This 360° view (events * level of expertise * relevant actors) over time will include the identification of complex situations where patients have a high need of expert care, and it will also highlight periods when the risk of coordination issues is increased.
* Compare care pathways depending on their referral to MSCU or not (before/after or here/elsewhere), with different kinds of outcomes (care trajectories, clinical parameters including therapies and MRI, as well as patient reported outcomes and experiences). Using indicators related to both objective and subjective health, MUSICALISE will help to understand the expected outcomes from MSCU, and how these structures contribute to improved experiences for people with MS and improved quality of care.

Our research question is "Under what conditions and how can the implementation of MSCU lead to better care integration and improved outcomes for people with MS and professionals according to their needs ?". This overarching question is declined into several sub-questions. What is the "ideal" care pathway according to people affected by MS and health care providers ? The hypothesis is that unmet needs regarding the appropriate care pathway and expectations regarding coordination may be different between patients and healthcare professionals, based on their respective experiences. In addition, it's expected that the level of expertise available in MSCU may not be necessary at every step throughout the disease course (phases of stable disease, good therapy responders, no specific health events...) nor feasible (time and costs constraints, human resources shortage). This would call for a model based upon "gradation of care" according to the needs of people with MS that optimizes referral to MSCU.

The aim will be to identify, with the patients, the coordination activities that punctuate patients' experience :

* Assessing all the needs and objectives of the patient and the professionals at the MSCU, including the patient's or carer's share of coordination ;
* Examine the development of the care plan and how it is personalised to the patient's unique circumstances and the role played by all the health and social care professionals involved ;
* Examine how the care plan is reviewed and updated as necessary ;
* Studying how care, medical and other appointments are planned ;
* Studying how care is provided directly to the patient ;
* Studying how the patient's state of health and needs are monitored and followed up (by the Expert Centre and locally) ;
* Studying how information is transferred between professionals and patients ;
* Studying how the patient is involved in the care pathway (involvement in decisions, collaboration with care providers) ;
* Studying the support methods used: therapeutic education, support for adherence to treatment, emotional support, technical support for monitoring biological parameters or carrying out administrative tasks, support from community resources, associations, etc.) ;
* Finally, studying how relational continuity is established by building a permanent, personal and meaningful relationship of mutual trust over time.

ELIGIBILITY:
Inclusion Criteria:

* Person diagnosed with MS;

  * Carer for someone with MS;
  * Healthcare professional working with MS patients;
  * Adult;
  * Person who has not objected to participating in the research.

Exclusion Criteria:

* Any person who has objected to the use of their data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: erson diagnosed with MS, carer for someone with MS, Healthcare professional working with MS patients.
Sampling Method: Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
most appropriate care pathway | Baseline
  In order to assess the care pathway as a whole, this survey will identify the key stages and characteristics that are likely to lead to a positive or negative experience of the care pathway. In order to define the most appropriate care pathway, proposals will be made, for example, on the most complex or risky moments in the pathway, the moments that require the greatest expertise in MS care.

CONTACTS AND LOCATIONS:
Locations (1):
- Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No